CLINICAL TRIAL: NCT06280885
Title: A Flexible Individualized ExeRcise Programme for Cancer Patients During ChEmotherapy
Acronym: FIERCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Emer Guinan, Associate Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FIERCE
Record Dates: First submitted 2023-12-06; First posted 2024-02-28 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Feasibility randomised controlled trial using a 2:1 randomisation
Masking Description: Not indicated for this feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIERCE Programme (Experimental): The FIERCE programme will consist of an aerobic and resistance exercise program delivered for the duration of chemotherapy.
  Exercise will be prescribed with the aim of achieving an overall exercise volume over the course of a chemotherapy cycle. The total volume of exercise prescribed in each cycle will be targeted towards achieving the exercise guidelines for cancer survivors which recommends 90 minutes of aerobic activity per week, in addition to resistance exercise at least two times per week.
  Exercise intensity will be autoregulated by participants based on how they are feeling on a given day. Participants will be given a choice of exercising at low, moderate, or higher intensity based on how BORG rating of perceived exertion (RPE) scale.
  Weekly check ins will be made to each participant over the phone by an exercise physiologist for goal setting. Participants will also be given a pedometer to monitor daily physical activity levels.
  Interventions: Behavioral: Exercise; Behavioral: Health Behaviour Change (Pedometer)
- Pedometer programme (Active Comparator): Participants randomized to the pedometer programme will receive individualised advice about exercising during chemotherapy and will also receive a pedometer to encourage daily activity. Participant in both groups will receive a personal exercise consultation to identify their individual needs and understand their exercise preferences.
  Interventions: Behavioral: Health Behaviour Change (Pedometer)

INTERVENTIONS:
Behavioral: Exercise — Participants will be randomised to either the FIERCE exercise programme involving supervised exercise prescription
  Arms: FIERCE Programme
Behavioral: Health Behaviour Change (Pedometer) — Participants in both arms will be provided with a pedometer as a health behaviour change intervention

SUMMARY:
The primary aim of this study is to measure the feasibility of delivering a co-designed exercise programme for patients with cancer receiving chemotherapy treatment.

DETAILED DESCRIPTION:
Exercise has been shown to play an important role in reducing many of the side effects associated with chemotherapy treatment. Exercise can help to improve symptoms of fatigue, nausea, muscle weakness, and pain, which in turn can help to improve patients overall quality of life and wellbeing. In addition to this, exercising during chemotherapy can also help to maintain physical fitness and preserve muscle mass, which has been shown to significantly reduce treatment toxicities. Despite these benefits of exercise, performing regular physical activity during chemotherapy poses significant challenges. Patients are faced with a number of physical and logistical barriers during chemotherapy which makes it difficult to engage in regular exercise. In addition to this, exercise programs that are being designed lack flexibility and individualization, and don't account for the unpredictable nature of chemotherapy treatment. It is, therefore, no surprise that patients struggle to meet the exercise recommendations during chemotherapy, and highlights the need for careful consideration when prescribing exercise during this time. In preparation for this study, the research team held a number of workshops which included a mixture of patients and healthcare professionals with the aim of co-designing an exercise intervention for patients during chemotherapy. Including public and patient involvement (PPI) in the design process will help to ensure that the exercise program that is developed is pragmatic and, most importantly, patient-centred.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18.
* Histological confirmed diagnosis of stage I to IIIc breast, ovarian or colorectal cancer.
* Scheduled to receive chemotherapy ± immunotherapy with curative intent.
* Medical clearance from oncologist to partake in regular exercise in accordance with American College of Sports Medicine (ACSM) preparticipation screening algorithm.
* Ability to provide written informed consent.

Exclusion Criteria:

* Advanced/metastatic disease.
* Scheduled to receive concurrent chemoradiotherapy.
* Scheduled to receive high-dose chemotherapy during hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment rates | At enrolement
  Recruitment rates will be calculated as the percentage of eligible participants who agreed to take part in the study. Recruitment rates will be calculated for each recruitment timepoint to determine which timepoint yields optimal recruitment. Reasons for declining recruitment will also be recorded.
Feasibility: Adherence rates | Through study completion, on average 6 months
  Exercise adherence will be used to measure the degree to which the participants performed the exercise at the desired intensity and time. After each exercise session, participants will be asked to rate their perceived exertion that they actually achieved during the exercise class. This RPE will be compared to the prespecified intensity that was chosen by the participant on the BORG scale at the beginning of the class to determine adherence to the intensity of the exercise session. Adherence to exercise time will be calculated by recording the total number of minutes spent exercising in each class compared to the total duration of the class.
Feasibility: Attendance rates | Through study completion, on average 6 months
  Exercise attendance will be calculated as the total number of exercise classes attended, either in-person or online, regardless of how much exercise was performed.
Feasibility: Retention Rates | Through study completion, on average 6 months
  Retention rates will be calculated as the number of participants who remained in the study at the end of the intervention as a proportion of the total number of participants recruited.
Feasibility: Reason for drop0out | Through study completion, on average 6 months
  Reasons for dropout will be recorded descriptively

SECONDARY OUTCOMES:
Cardiorespiratory Fitness | Pre and post intervention (on average 6 months)
  Cardiorespiratory fitness will be estimated using the submaximal Astrand-Rhyming Cycle Ergometer Test (ARCET). The test will be performed on a cycle ergometer and will include breath-by-breath analysis using COSMED QUARK equipment.
Muscular Strength | Pre and Post intervention, on average 6 months
  Leg Strength Leg strength will be measured using a 1 repetition max (1RM) leg press test. Participants will complete a warm-up of 6 repetitions at approximately 60% 1RM followed by 3 repetitions at 80% 1RM. Following successful completion of the warm-up repetitions, participants will perform a maximum effort to determine their 1RM. Participants will be given a maximum of 5 attempts to determine their 1RM with a 2-minute rest between each attempt.
  Hand Grip Strength Hand grip strength (HGS) will be measured using a hand-held dynamometer. Participants will perform the test in a seated position, with their elbow at 90 degrees. Participants will be instructed to squeeze on the handle using maximum effort for 3 seconds. Three attempts will be made on each hand with a 1-minute rest between attempts. The highest value will be recorded.
Body Mass Index | Pre and Post intervention, on average 6 months
  Weight (kilogrammes (kg)) and height (centimetres (cm)) will be recorded by standard methods using a calibrated scales and stadiometer. Body mass index (BMI) will be calculated as weight (kg)/ height (metres (m2)).
Mid-arm circumference | Pre and Post intervention, on average 6 months
  Mid-arm muscle circumference will be measured in centimetres at the halfway point between the olecranon process of the ulna and the acromion process of the scapula.
Waist Circumference | Pre and Post intervention, on average 6 months
  Waist circumference will be measured in centimetres at the mid-point between the iliac crest and the 12th rib following gentle expiration. Circumferential measurements will be taken in duplicate and averaged for data entry.
Bioimpedance Analysis | Pre and Post intervention, on average 6 months
  Bioimpedance analysis (BIA) will be used to determine body composition and will be performed using the SECA mBCA 515 (Seca, Hamburg, Germany). Measures recorded will include; fat mass, fat free mass, and skeletal muscle mass (all measured in kg).
Health Related Quality of Life | Pre and Post intervention, on average 6 months
  Health-related quality of life will be determined by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30 version 3.0). This validated instrument assessed quality of life in functional, symptom and global domains. Scores for each question were calculated according to the EORTC QLQ-C30 manual and linearly transformed into a 0-100 scale A high score for a functional scale indicates a high level of functioning. A high score for a symptom scale/single item represents a high symptom burden.
Fatigue | Pre and Post intervention, on average 6 months
  Fatigue will be measured using the Cancer Fatigue Scale (CFS). The CFS is a 15-item scale comprising of 3 subscales, physical (maximum score 28), affective (maximum score 16), and cognitive (maximum score 16), with a total score range from 0-60. Higher scores reveal more severe fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- St James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kearney N, Connolly D, Bahramian K, Sheill G, Coghlan-Lynch K, O'Sullivan J, Coleman N, O'Hanlon Brown C, Gallagher D, O'Gorman C, O'Brien C, Tierney A, Rankin K, O'Neill L, Guinan E. A Flexible Individualised ExeRcise programme for cancer patients during ChEmotherapy (FIERCE): Protocol for a randomised controlled feasibility trial. Contemp Clin Trials. 2025 Jun;153:107923. doi: 10.1016/j.cct.2025.107923. Epub 2025 Apr 21. PMID 40268238